CLINICAL TRIAL: NCT03632473
Title: Validation of Multimodal Evoked Potentials (mmEP) for Predicting Disease Progression in Multiple Sclerosis: Sub-study Within the Swiss Multiple Sclerosis Cohort (SMSC)
Brief Title: Validation of Multimodal Evoked Potentials (mmEP) for Predicting Disease Progression in Multiple Sclerosis
Acronym: SMSC
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01818; me14Fuhr
Record Dates: First submitted 2018-07-26; First posted 2018-08-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Multiple Sclerosis
Keywords: Multimodal Evoked potentials; Visual evoked potentials; Somato-sensory evoked potentials; Motor evoked potentials; Expanded Disability Status Scale (EDSS)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- clinically isolated syndrome (CIS): Multiple sclerosis (MS) with a clinically isolated syndrome (CIS) within six months of first clinical event.
  Multimodal evoked potentials (mmEP) assessments will take place at baseline, month 12 (from baseline), month 24 (from baseline) and month 36 (from baseline)
  Interventions: Diagnostic Test: multimodal evoked potentials (mmEP)
- early relapsing-remitting late disease course (RRMS): MS with relapsing-remitting early disease course (RRMS) </= 10 years, Expanded Disability Status Scale (EDSS) </=3.5
  EDSS:
  1.0: No disability, minimal signs in 1 functional System (FS) 1.5: No disability, minimal signs in more than one FS 2.0: Minimal disability in one FS 2.5: Mild disability in one FS or minimal disability in two FS 3.0: Moderate disability in one FS, or mild disability in three or four FS. No impairment to Walking 3.5: Moderate disability in one FS and more than minimal disability in several others. No impairment to Walking.
  Multimodal evoked potentials (mmEP) assessments will take place at baseline, month 12 (from baseline), month 24 (from baseline) and month 36 (from baseline)
  Interventions: Diagnostic Test: multimodal evoked potentials (mmEP)
- late relapsing-remitting late disease course (RRMS): MS with relapsing-remitting late disease course (late RRMS) of 5 to 15 years, EDSS: 2.0-5.5 inclusive
  EDSS:
  4.0: Significant disability but self-sufficient and up and about some 12 hours a day. Able to walk without aid or rest for 500m 4.5: Significant disability but up and about much of the day, able to work a full day, may otherwise have some limitation of full activity or require minimal assistance. Able to walk without aid or rest for 300m 5.0: Disability severe enough to impair full daily activities and ability to work a full day without special provisions. Able to walk without aid or rest for 200m 5.5: Disability severe enough to preclude full daily activities. Able to walk without aid or rest for 100m.
  Multimodal evoked potentials (mmEP) assessments will take place at baseline, month 12 (from baseline), month 24 (from baseline) and month 36 (from baseline)
  Interventions: Diagnostic Test: multimodal evoked potentials (mmEP)
- primary progressive disease course (PPMS): MS with a primary progressive disease course (PPMS) up to 15 years, EDSS: 2.0-6.5 inclusive
  EDSS:
  6.0: Requires a walking aid - cane, crutch, etc. - to walk about 100m with or without resting 6.5: Requires two walking aids - pair of canes, crutches, etc. - to walk about 20m without resting.
  Multimodal evoked potentials (mmEP) assessments will take place at baseline, month 12 (from baseline), month 24 (from baseline) and month 36 (from baseline)
  Interventions: Diagnostic Test: multimodal evoked potentials (mmEP)

INTERVENTIONS:
Diagnostic Test: multimodal evoked potentials (mmEP) — combination of visual evoked potentials (VEP) and motor evoked potentials (MEP) or the combination of VEP, MEP and somato-sensory evoked potentials (SSEP)

SUMMARY:
Utility of Multimodal Evoked potentials (mmEP) for monitoring disease course and prediction of progression at different stages of Multiple Sclerosis (MS) is investigated

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with a clinically isolated syndrome (CIS) or MS with a relapsing-remitting (RRMS) or a primary progressive disease course (PPMS):
* CIS: EDSS <= 5.5 within six months of first clinical event
* early RRMS: EDSS: <= 3.5 disease course of 5 up to 10 years
* late RRMS: EDSS: 2.0-5.5 inclusive disease course of 5 to 15 years
* PPMS: EDSS: 2.0-6.5 inclusive disease course up to 15 years
* participation in the Swiss Multiple Sclerosis Cohort Study (SMSC)
* mental ability to cooperate
* written informed consent

Exclusion Criteria:

* alcohol or substance abuse
* progressive disease other than Multiple Sclerosis
* psychiatric disorder requiring a treatment by a psychiatrist
* patients with movable metal implants, e.g. pace-maker, stents, deep brain stimulators etc.;(patients with jaw- or bone-fixed metal implants can be included)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MS patients participating in the Swiss Multiple Sclerosis Cohort Study (SMSC), regardless of MS-specific treatment
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
correlation of EP-sum-score (Σ-EP) and the Expanded Disability Status Scale (EDSS) | 3 years
  logistic regression model will be used to predict worsening in EDSS defined by a 1-point-change (0.5 if EDSS is 5.5 or higher) at year 3

CONTACTS AND LOCATIONS:
Overall Officials: Peter Fuhr, Prof., Principal Investigator — Dep. of Neurology, Hospital of the University of Basel
Locations (3):
- Switzerland (3):
  - Dep. of Neurology, Hospital of the University of Basel, Basel
  - Hopitaux universitaires de Genève, Geneva
  - Neurocenter of Southern Switzerland, Ospedale Regionale di Lugano, Lugano

REFERENCES:
- [Background] Hardmeier M, Schlaeger R, Lascano AM, Toffolet L, Schindler C, Gobbi C, Lalive P, Kuhle J, Kappos L, Fuhr P. Prognostic biomarkers in primary progressive multiple sclerosis: Validating and scrutinizing multimodal evoked potentials. Clin Neurophysiol. 2022 May;137:152-158. doi: 10.1016/j.clinph.2022.02.019. Epub 2022 Mar 7. PMID 35316624
- [Background] Hardmeier M, Fuhr P. Multimodal Evoked Potentials as Candidate Prognostic and Response Biomarkers in Clinical Trials of Multiple Sclerosis. J Clin Neurophysiol. 2021 May 1;38(3):171-180. doi: 10.1097/WNP.0000000000000723. PMID 33958567
- [Background] Hardmeier M, Schindler C, Kuhle J, Fuhr P. Validation of Quantitative Scores Derived From Motor Evoked Potentials in the Assessment of Primary Progressive Multiple Sclerosis: A Longitudinal Study. Front Neurol. 2020 Jul 24;11:735. doi: 10.3389/fneur.2020.00735. eCollection 2020. PMID 32793104
- [Background] Hardmeier M, Jacques F, Albrecht P, Bousleiman H, Schindler C, Leocani L, Fuhr P. Multicentre assessment of motor and sensory evoked potentials in multiple sclerosis: reliability and implications for clinical trials. Mult Scler J Exp Transl Clin. 2019 May 1;5(2):2055217319844796. doi: 10.1177/2055217319844796. eCollection 2019 Apr-Jun. PMID 31069107